CLINICAL TRIAL: NCT01857063
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled Cross-over Clinical Trial to Study the Efficacy and Safety of MK-0476 in Japanese Pediatric Subjects With Seasonal Allergic Rhinitis
Brief Title: Study of the Efficacy and Safety of MK-0476 in Japanese Pediatric Participants With Seasonal Allergic Rhinitis (MK-0476-519)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0476-519; 132232 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast/Placebo (Experimental): Participants receive montelukast 5 mg chewable tablets for 7 days during Period 1 and receive placebo chewable tablets for 7 days during Period 2. There is a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: Montelukast; Drug: Placebo
- Placebo/Montelukast (Experimental): Participants receive placebo chewable tablets for 7 days during Period 1 and receive montelukast 5 mg chewable tablets for 7 days during Period 2. There is a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: Montelukast; Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast 5 mg chewable tablets, taken orally once daily at bedtime for 7 days
  Other Names: montelukast sodium
Drug: Placebo — Matching placebo chewable tablets, taken orally once daily at bedtime for 7 days

SUMMARY:
This study will evaluate the efficacy and safety of montelukast (MK-0476) in the treatment of Japanese pediatric participants with seasonal allergic rhinitis (SAR). The primary hypothesis of this study is that montelukast is superior to placebo in the treatment of nasal symptoms in SAR.

ELIGIBILITY:
Inclusion Criteria:

* Weight: ≥ 25 kg
* Height: ≥ 125 cm
* Able to record symptoms in a diary
* Has had allergic rhinitis symptoms [Japanese Cedar (JC) pollinosis]
* Tested positive for JC pollen specific immunoglobulin E (IgE) antibody assay

Exclusion Criteria:

* Has nasal findings that would interfere with evaluating nasal congestion symptoms
* Past or present medical history of bronchial asthma
* Medical history of allergies except allergic rhinitis and has possibility of dramatically worsening of these symptoms induced by JC pollen exposure

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2013-09-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hashiguchi K, Okubo K, Inoue Y, Numaguchi H, Tanaka K, Oshima N, Mehta A, Nishida C, Saito I, Philip G. Evaluation of Montelukast for the Treatment of Children With Japanese Cedar Pollinosis Using an Artificial Exposure Chamber (OHIO Chamber). Allergy Rhinol (Providence). 2018 Jul 13;9:2152656718783599. doi: 10.1177/2152656718783599. eCollection 2018 Jan-Dec. PMID 30027002

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (7 Days)
Arm/Group | Montelukast/Placebo | Placebo/Montelukast
Started | 110 | 110
Completed | 108 | 106
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Period: Period 2 (7 Days)
Arm/Group | Montelukast/Placebo | Placebo/Montelukast
Started | 108 | 106
Completed | 104 | 104
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast/Placebo | Placebo/Montelukast | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (1.6) [10 to 15] | 12.7 (1.5) [10 to 15] | 12.5 (1.6) [10 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 59 | 114
  Male | 55 | 51 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Averaged During 3 Hours of Exposure
Description: The TNSS is the sum of the three nasal symptom scores for nasal congestion, nasal discharge and sneezing. Participants completed a questionnaire about their nasal symptoms. Score ranged from 0 to 4 for each of the three nasal symptoms, with a total possible score ranging from 0 to 12 and a higher score indicating more severe nasal symptoms. The baseline TNSS was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline TNSS was assessed on Day 7 of a treatment period during 3 hours of exposure to Japanes cedar (JC) pollen in the chamber room, as an average of measurements at 30, 60, 90, 120, 150 and 180 minutes. Analysis was done by study drug as taken.
Time Frame: Baseline and after 3 hours of pollen exposure on Day 7 of each treatment period
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who took at least one dose of study drug, and had a baseline assessment and at least one post-baseline assessment in a treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Montelukast: Participants receive montelukast 5 mg for 7 days, regardless of sequence.
- Placebo: Participants receive placebo for 7 days, regardless of sequence.
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale | 1.17 [1.03 to 1.31] | 1.18 [1.04 to 1.32]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.913, Longitudinal Data Analysis (LDA) — Longitudinal Data Analysis (LDA) model with baseline TNSS as a covariate, sequence, treatment and period as fixed effects and participant as a random effect; Difference in Least Squares (LS) Means = -0.01, 95% CI 2-sided [-0.11 to 0.10]

2. Primary Outcome: Percentage of Participants Who Experience at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Participants were monitored for occurrence adverse events for up to 14 days after last dose of study drug. Analysis was done by study drug as taken.
Time Frame: Up to 5 weeks
Population: The All Patients as Treated (APaT) population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 216 | 218
percentage of participants | 10.2 | 16.5

3. Secondary Outcome: Change From Baseline in Weighted TNSS Averaged During 3 Hours of Exposure
Description: TNSS was weighted as 2:1:1 for nasal congestion, nasal discharge and sneezing. The Weighted TNSS ranged from 0 to 16, with a higher score indicating more severe weighted total nasal symptoms. The baseline Weighted TNSS was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline TNSS was assessed on Day 7 of a treatment period during 3 hours of exposure to JC pollen in the chamber room, as an average of measurements at 30, 60, 90, 120, 150 and 180 minutes. Analysis was done by study drug as taken.
Time Frame: Baseline and after 3 hours of pollen exposure on Day 7 of each treatment period
Population: The FAS population consisted of all randomized participants who took at least one dose of study drug, and had a baseline assessment and at least one post-baseline assessment in a treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale | 1.85 [1.63 to 2.07] | 1.86 [1.63 to 2.08]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.953, LDA — Longitudinal Data Analysis (LDA) model with baseline Weighted TNSS as a covariate, sequence, treatment and period as fixed effects and participant as a random effect; Difference in LS Means = -0.00, 95% CI 2-sided [-0.17 to 0.16]

4. Secondary Outcome: Change From Baseline in Nasal Congestion Score Averaged During 3 Hours of Exposure
Description: The Nasal Congestion Score was assessed as 0 = No symptoms of nasal congestion to 4 = Completely obstructed all day, with a possible Nasal Congestion Score ranging from 0 to 4 and a higher score indicating more severe nasal congestion. The baseline Nasal Congestion Score was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline Nasal Congestion Score was assessed on Day 7 of a treatment period during 3 hours of exposure to JC pollen in the chamber room, as an average of measurements at 30, 60, 90, 120, 150 and 180 minutes. Analysis was done by study drug as taken.
Time Frame: Baseline and after 3 hours of pollen exposure on Day 7 of each treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale | 0.68 [0.59 to 0.76] | 0.68 [0.59 to 0.76]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.974, LDA — Longitudinal Data Analysis (LDA) model with baseline nasal congestion score as a covariate, sequence, treatment and period as fixed effects and participant as a random effect; Difference in LS Means = -0.00, 95% CI 2-sided [-0.07 to 0.07]

5. Secondary Outcome: Change From Baseline in Nasal Discharge Score Averaged During 3 Hours of Exposure
Description: The Nasal Discharge Score was assessed as 0 = 0 times participant blew his/her nose to 4 = 21 or more times participant blew his/her nose, with a possible Nasal Discharge Score ranging from 0 to 4 and a higher score indicating more severe nasal discharge. The baseline Nasal Discharge Score was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline Nasal Discharge Score was assessed on Day 7 of a treatment period during 3 hours of exposure to JC pollen in the chamber room, as an average of measurements at 30, 60, 90, 120, 150 and 180 minutes. Analysis was done by study drug as taken.
Time Frame: Baseline and after 3 hours of pollen exposure on Day 7 of each treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale | 0.29 [0.25 to 0.34] | 0.32 [0.27 to 0.37]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.182, LDA — Longitudinal Data Analysis (LDA) model with baseline nasal discharge score as a covariate, sequence, treatment and period as fixed effects and participant as a random effect; Difference in LS Means = -0.03, 95% CI 2-sided [-0.06 to 0.01]

6. Secondary Outcome: Change From Baseline in Sneezing Score Averaged During 3 Hours of Exposure
Description: The Sneezing Score was assessed as 0 = 0 times participant sneezed to 4 = 21 or more times participant sneezed, with a possible Sneezing Score ranging from 0 to 4 and a higher score indicating more severe sneezing. The baseline Sneezing Score was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline Sneezing Score was assessed on Day 7 of a treatment period during 3 hours of exposure to JC pollen in the chamber room, as an average of measurements at 30, 60, 90, 120, 150 and 180 minutes. Analysis was done by study drug as taken.
Time Frame: Baseline and after 3 hours of pollen exposure on Day 7 of each treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale | 0.20 [0.16 to 0.24] | 0.18 [0.14 to 0.22]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.161, LDA — Longitudinal Data Analysis (LDA) model with baseline sneezing score as a covariate, sequence, treatment and period as fixed effects and participant as a random effect; Difference in LS Means = 0.02, 95% CI 2-sided [-0.01 to 0.05]

7. Secondary Outcome: Change From Baseline in TNSS at 30, 60, 90, 120, 150 and 180 Minutes After Entering Chamber Room
Description: The TNSS is the sum of the three nasal symptom scores for nasal congestion, nasal discharge and sneezing. The possible TNSS ranged from 0 to 12, with a higher score indicting more severe total nasal symptoms. The baseline TNSS was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline TNSS was assessed on Day 7 of a treatment period at 30, 60, 90, 120, 150 and 180 minutes after entering the chamber room. Analysis was done by study drug as taken.
Time Frame: Baseline and at 30, 60, 90, 120, 150 and 180 minutes after entering chamber room on Day 7 of a treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale
  30 minutes after entering chamber room | 0.54 [0.42 to 0.67] | 0.59 [0.46 to 0.71]
  60 minutes after entering chamber room | 1.00 [0.84 to 1.16] | 1.07 [0.91 to 1.23]
  90 minutes after entering chamber room | 1.36 [1.18 to 1.55] | 1.31 [1.12 to 1.49]
  120 minutes after entering chamber room | 1.38 [1.18 to 1.57] | 1.35 [1.16 to 1.54]
  150 minutes after entering chamber room | 1.38 [1.19 to 1.57] | 1.35 [1.16 to 1.54]
  180 minutes after entering chamber room | 1.39 [1.19 to 1.59] | 1.40 [1.21 to 1.60]

8. Secondary Outcome: Change From Baseline in Weighted TNSS at 30, 60, 90, 120, 150 and 180 Minutes After Entering Chamber Room
Description: TNSS was weighted as 2:1:1 for nasal congestion, nasal discharge and sneezing. The possible Weighted TNSS ranged from 0 to 16, with a higher score indicating more severe total nasal symptoms. The baseline TNSS was assessed on Day 7 of a treatment period prior to entering the chamber room. The post-baseline Weighted TNSS was assessed on Day 7 of a treatment period at 30, 60, 90, 120, 150 and 180 minutes after entering the chamber room. Analysis was done by study drug as taken.
Time Frame: Baseline and at 30, 60, 90, 120, 150 and 180 minutes after entering chamber room on Day 7 of a treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale
  30 minutes after entering chamber room | 0.86 [0.67 to 1.05] | 0.91 [0.72 to 1.11]
  60 minutes after entering chamber room | 1.55 [1.31 to 1.79] | 1.63 [1.40 to 1.87]
  90 minutes after entering chamber room | 2.11 [1.83 to 2.38] | 2.04 [1.76 to 2.32]
  120 minutes after entering chamber room | 2.17 [1.87 to 2.47] | 2.17 [1.87 to 2.47]
  150 minutes after entering chamber room | 2.21 [1.92 to 2.51] | 2.16 [1.86 to 2.46]
  180 minutes after entering chamber room | 2.22 [1.91 to 2.53] | 2.21 [1.90 to 2.52]

9. Secondary Outcome: Change From Baseline in Nasal Congestion Score at 30, 60, 90, 120, 150 and 180 Minutes After Entering Chamber Room
Description: The Nasal Congestion Score was assessed as 0 = No symptoms of nasal congestion to 4 = Completely obstructed all day. The possible Nasal Congestion Score ranged from 0 to 4, with a higher score indicating more severe nasal congestion.The Nasal Congestion Score was assessed on Day 7 prior to entering the chamber room and at 30, 60, 90, 120, 150 and 180 minutes after entering the chamber room. Analysis was done by study drug as taken.
Time Frame: Baseline and at 30, 60, 90, 120, 150 and 180 minutes after entering chamber room on Day 7 of a treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale
  30 minutes after entering chamber room | 0.32 [0.24 to 0.39] | 0.33 [0.25 to 0.40]
  60 minutes after entering chamber room | 0.55 [0.46 to 0.63] | 0.56 [0.48 to 0.65]
  90 minutes after entering chamber room | 0.74 [0.64 to 0.85] | 0.73 [0.63 to 0.83]
  120 minutes after entering chamber room | 0.80 [0.68 to 0.91] | 0.82 [0.70 to 0.94]
  150 minutes after entering chamber room | 0.83 [0.72 to 0.95] | 0.81 [0.70 to 0.93]
  180 minutes after entering chamber room | 0.83 [0.70 to 0.95] | 0.81 [0.69 to 0.93]

10. Secondary Outcome: Change From Baseline in Nasal Discharge Score at 30, 60, 90, 120, 150 and 180 Minutes After Entering Chamber Room
Description: The Nasal Discharge Score was assessed as 0 = 0 times participant blew his/her nose to 4 = 21 or more times participant blew his/her nose. The possible Nasal Discharge Score ranged from 0 to 4, with a higher score indicating more severe nasal discharge.The Nasal Discharge Score was assessed on Day 7 prior to entering the chamber room and at 30, 60, 90, 120, 150 and 180 minutes after entering the chamber room. Analysis was done by study drug as taken.
Time Frame: Baseline and at 30, 60, 90, 120, 150 and 180 minutes after entering chamber room on Day 7 of a treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale
  30 minutes after entering chamber room | 0.13 [0.08 to 0.18] | 0.17 [0.12 to 0.22]
  60 minutes after entering chamber room | 0.27 [0.21 to 0.34] | 0.33 [0.27 to 0.40]
  90 minutes after entering chamber room | 0.39 [0.32 to 0.46] | 0.38 [0.31 to 0.45]
  120 minutes after entering chamber room | 0.34 [0.27 to 0.40] | 0.36 [0.29 to 0.42]
  150 minutes after entering chamber room | 0.31 [0.24 to 0.37] | 0.32 [0.25 to 0.39]
  180 minutes after entering chamber room | 0.33 [0.26 to 0.40] | 0.37 [0.30 to 0.44]

11. Secondary Outcome: Change From Baseline in Sneezing Score at 30, 60, 90, 120, 150 and 180 Minutes After Entering Chamber Room
Description: The Sneezing Score was assessed as 0 = 0 times participant sneezed to 4 = 21 or more times participant sneezed. The possible Sneezing Score ranged from 0 to 4, with a higher score indicating more severe sneezing. The Sneezing Score was assessed on Day 7 prior to entering the chamber room and at 30, 60, 90, 120, 150 and 180 minutes after entering the chamber room. Analysis was done by study drug as taken.
Time Frame: Baseline and at 30, 60, 90, 120, 150 and 180 minutes after entering chamber room on Day 7 of a treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 213 | 211
score on a scale
  30 minutes after entering chamber room | 0.09 [0.05 to 0.14] | 0.09 [0.05 to 0.14]
  60 minutes after entering chamber room | 0.18 [0.12 to 0.23] | 0.18 [0.12 to 0.23]
  90 minutes after entering chamber room | 0.23 [0.16 to 0.29] | 0.20 [0.13 to 0.26]
  120 minutes after entering chamber room | 0.25 [0.19 to 0.31] | 0.17 [0.11 to 0.23]
  150 minutes after entering chamber room | 0.24 [0.18 to 0.30] | 0.21 [0.15 to 0.27]
  180 minutes after entering chamber room | 0.23 [0.17 to 0.30] | 0.23 [0.16 to 0.29]

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug (Up to 5 weeks)
Description: The All Patients as Treated (APaT) population consisted of all randomized participants who received at least one dose of study drug.
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/218
Other Adverse Events (participants affected / at risk) | 10/216 | 17/218
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=216) | Placebo (N=218)
Protein urine present (Investigations) | 10 (10) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.